CLINICAL TRIAL: NCT00961311
Title: Evaluation of Acute Safety and Efficacy of the Medtronic Sprinter Legend 1.25mm Balloon Dilation Catheter Utilized for Enlarging Coronary Luminal Diameters During PCI Procedures
Brief Title: Sprinter Legend Balloon Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-111
Record Dates: First submitted 2009-07-14; First posted 2009-08-18 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Balloon; Angioplasty; Coronary Artery; PCI; PTCA; Heart Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trial Arm (Experimental): All patients with systematic ischemic heart disease with stenotic lesions that are amenable to percutaneous treatment.
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: Sprinter Legend 1.25mm Balloon Catheter

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Balloon angioplasty of a severely stenotic coronary lesion with the Sprinter Legend 1.25mm Balloon.
Device: Sprinter Legend 1.25mm Balloon Catheter — Balloon Angioplasty

SUMMARY:
Open label, single-arm trial to study the safety and effectiveness of the Sprinter Legend 1.25 mm angioplasty balloon.

DETAILED DESCRIPTION:
The study examines acute outcomes when the Sprinter Legend 1.25mm balloon catheter is used for enlarging coronary luminal diameters during PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than18 years of age and able to give informed consent.
* Patient with stenotic lesions in coronary arteries or bypass graft stenosis that are suitable for percutaneous coronary intervention (PCI).
* The patient has single or multiple vessel coronary artery disease and clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, and/or a positive functional study.
* Female patients of childbearing potential must have a negative pregnancy test within seven (7) days before the procedure.
* Patient or patient's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective investigational site.
* Patients with symptomatic ischemic heart disease due to stenotic lesions in coronary arteries or bypass graft stenosis that are amenable to percutaneous treatment.

Exclusion Criteria:

* A known hypersensitivity or contraindication to aspirin, heparin, or bivalirudin, anti-platelet medications, or sensitivity to contrast media, which cannot be adequately pre-medicated.
* A serum creatinine level > 2.0 mg/dl within seven days prior to index procedure.
* Evidence of an acute myocardial infarction within 72 hours of the intended index procedure (defined as: Q wave myocardial infarction or non-Q wave myocardial infarction having creatine kinase myocardial-band isoenzyme (CK-MB) or troponin elevated above the Institution's upper limit of normal).
* During the index procedure, the target lesion requires additional treatment with a cutting balloon, any artherectomy, any laser, thrombectomy, etc.
* History of stroke or transient ischemic attack (TIA) within the prior 6 months.
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Scripps Green Hospital
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States

REFERENCES:
- [Result] Kandzari DE, Zankar AA, Teirstein PS, Brilakis ES, Banerjee S, Price MJ, Stinis CT, Hudson PA, Dahle TG, Eng M, Brown R, Ferguson A, Addo TA, Popma JJ. Clinical outcomes following predilation with a novel 1.25-mm diameter angioplasty catheter. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):510-4. doi: 10.1002/ccd.22734. Epub 2010 Nov 4. PMID 21351225

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Angioplasty: All patients with systematic ischemic heart disease with stenotic lesions that are amenable to percutaneous coronary treatment. Study participants were treated with the Sprinter Legend 1.25mm angioplasty balloon.
Period: Overall Study
Arm/Group | Balloon Angioplasty
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Angioplasty
Number analyzed (Participants) | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: Procedural Success defined as delivery of the balloon to the target lesion, no evidence of perforation or dissection and restoration of normal blood flow at the end of the procedure.
Time Frame: 1-3 days
Measure: Number; unit: Percent of Participants
Arm/Group | Balloon Angioplasty
Number analyzed (Participants) | 51
Percent of Participants | 100

2. Secondary Outcome: Major Adverse Cardic Events (MACE)
Description: Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction, emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods.
Time Frame: 1-3 days
Measure: Number; unit: Percent of Participants
Arm/Group | Balloon Angioplasty
Number analyzed (Participants) | 51
Percent of Participants | 2.0

3. Secondary Outcome: Vessel Perforation (Clinical)
Description: Clinical vessel perforation is classified as requring additional treatment, or resulting in significant pericardial effusion, acute closure, myocardial infarction, or death.
Time Frame: 1-3 days
Measure: Number; unit: Percent of Participants
Arm/Group | Balloon Angioplasty
Number analyzed (Participants) | 51
Percent of Participants | 0

4. Secondary Outcome: Device Success
Description: Device Success defined as successful delivery of the balloon to the target lesion, dilatation of the lesion using the study device, and no evidence of arterial perforation, dissection, arrhythmias, or reduction in blood flow.
Time Frame: 1-3 days
Measure: Number; unit: Percent of Participants
Arm/Group | Balloon Angioplasty
Number analyzed (Participants) | 51
Percent of Participants | 100

ADVERSE EVENTS:
Time Frame: 1-3 days
Arm/Group | Balloon Angioplasty
Serious Adverse Events (participants affected / at risk) | 6/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Angioplasty (N=51)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Cardiac Enzymes Increased (Investigations) | 3 (3)
Renal Failure (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and or Participating lnstitution may publish the results of work performed in accordance with the Publication Strategy described in the Clinical Investigational Plan; provided, however, that any such publication or presentation shall be at a time determined by Medtronic and shall be provided to Medtronic for review at least 60 days prior to submission or presentation, for a determination by Medtronic of whether Confidential lnformation is disclosed.